CLINICAL TRIAL: NCT00105404
Title: A Randomized Trial Comparing Intravitreal Triamcinolone Acetonide and Laser Photocoagulation for Diabetic Macular Edema
Brief Title: Treatment of Diabetic Macular Edema: Triamcinolone Injections Vs. Laser Photocoagulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050107; 05-EI-0107
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-10-30

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; DME
Keywords: Steroid; Diabetic Macular Edema; DME
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide

SUMMARY:
This study will compare the side effects of two treatments for diabetic macular edema, in which blood vessels in the retina (tissue that lines the back of the eye) become leaky and the retina and macula (the center part of the retina that is responsible for fine vision) swell, causing vision loss.

Patients 18 years of age and older with diabetes mellitus and macular edema in one or both eyes may be eligible for this study. Candidates are screened with the following tests and procedures:

* Blood pressure measurement.
* Blood tests to measure HbA1c, a measure of the patient's diabetes control.
* Eye examination to assess visual acuity and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils are dilated with drops for this examination.
* Eye photography to help evaluate the status of the retina and changes that may occur in the future. Photographs of the inside of the eye are taken using a camera that flashes a bright light into the eye.
* Electroretinograms (ERG) to measure electrical responses generated in the retina. Wearing eye patches, the patient sits in a dark room for 30 minutes. Then, electrodes are taped to the forehead and an earlobe. The eye patches are removed, the surface of the eye is numbed with eye drops, and contact lenses are placed on the eyes. The patient looks inside a white globe that emits a series of light flashes for about 20 minutes. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Optical coherence tomography to measure retinal thickness. The eye is examined with a machine that produces cross-sectional pictures of the retina. These measurements are repeated during the study to determine whether retinal thickening is improving, worsening, or staying the same.

Patients with macular edema in both eyes receive laser therapy in one eye and triamcinolone injections in the other. Patients with just one affected eye are randomly assigned to receive either laser or triamcinolone treatment. Those who receive only laser therapy may later receive triamcinolone injections in the second eye if it, too, develops macular edema.

For the laser treatment, the eye surface is numbed with drops and a contact lens is placed on the eye during the laser beam application. Before the treatment, patients may have fluorescein angiography, in which pictures of the retina are taken using a yellow dye. The dye is injected into a vein and travels to the blood vessels in the eye. The camera flashes a blue light in the eye and takes pictures that show the amount of dye leakage into the retina. This helps guide the laser treatment. Patients return for follow-up visits every 4 months for 3 years. If the macular edema is gone, no additional treatment is given and patients are followed as often as every 2 months. If the edema does return, additional treatments may be done at subsequent visits. Patients whose vision worsens considerably at the end of 1 year may be treated with a steroid injection, unless the other eye has also been treated with triamcinolone.

For the triamcinolone injections, numbing drops, antibiotic drops, and drops to dilate the pupil, and possibly and anesthetic injection, are put in the eye before the medicine is injected into the vitreous (jelly-like substance inside the eye). Then, the patient lies on his or her back for 30 minutes before being discharged home. Patients return for follow-up visits 4 days and 4 weeks after the injection, and then every 4 months for 3 years. Patients whose edema resolves are followed as often as every 2 months. Those whose edema returns have additional injections at the 4-month visits. Patients whose condition does not improve after 1 year or whose vision worsens may undergo laser treatment.

DETAILED DESCRIPTION:
Diabetic retinopathy is a major cause of visual impairment in the United States. Diabetic Macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20% in patients with type 1 diabetes mellitus (DM), 25% in patients with type 2 DM who are taking insulin, and 14% in patients with type 2 DM who do not take insulin.

In a review of three early studies concerning the natural history of diabetic macular edema, Ferris and Patz found that 53% of 135 eyes with diabetic macular edema, presumably all involving the center of the macula, lost two or more lines of visual acuity over a two year period. In the Early Treatment Diabetic Retinopathy Study (ETDRS), 33% of 221 untreated eyes available for follow-up at the 3-year visit, all with edema involving the center of the macula at baseline, had experienced a 15 or more letter decrease in visual acuity score (equivalent to a doubling of the visual angle, e.g., 20/25 to 20/50, and termed moderate visual loss).

The frequency of an unsatisfactory outcome following laser photocoagulation in some eyes with diabetic macular edema has prompted interest in other treatment modalities. One such treatment is pars plana vitrectomy. These studies suggest that vitreomacular traction, or the vitreous itself, may play a role in increased retinal vascular permeability. Removal of the vitreous or relief of mechanical traction with vitrectomy and membrane stripping may be followed by substantial resolution of macular edema and corresponding improvement in visual acuity. However, this treatment may be applicable only to a specific subset of eyes with diabetic macular edema. It also requires a complex surgical intervention with its inherent risks, recovery time, and expense. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors and antibodies targeted at vascular endothelial growth factor (VEGF) are under investigation. The use of intravitreal corticosteroids is another treatment modality that has generated recent interest.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

(Subject-Level Inclusion Criteria:)

To be eligible, the following inclusion criteria (1-6) must be met:

1. Age greater than or equal to 18 years.
2. Diagnosis of diabetes mellitus (type 1 or type 2).

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   * Current regular use of insulin for the treatment of diabetes
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   * Documented diabetes by ADA and/or WHO criteria
3. At least one eye meets the study eye criteria.
4. If only one eye eligible, fellow eye meets criteria
5. Able and willing to provide informed consent.
6. Patient understands that (1) if both eyes are eligible at the time of randomization, one eye will receive intravitreal triamcinolone ancetonide and one eye will receive laser, and (2) if only one eye is eligible at the time of randomization and the fellow eye develops DME later, then the fellow eye will not receive intravitreal triamcinolone ancetonide if the study eye received intravitreal triamcinolone ancetonide (however, if the study eye was assigned to the laser group, then the fellow eye may be treated with the 4mg dose of the study intravitreal triamcinolone ancetonide formulation, provided the eye assigned to laser has not received an intravitreal injection; such an eye will not be a study eye but since it is receiving study drug, it will be followed for adverse effects).

   (Subject-Level Exclusion Criteria:)

   A patient is not eligible if any of the following exclusion criteria (7-13) are present:
7. History of chronic renal failure requiring dialysis or kidney transplant.
8. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

   - Patients in poor gylcemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
9. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.
10. Known allergy to any corticosteroid or any component of the delivery vehicle.
11. History of systemic (e.g., oral, IV, IM, epidural, bursal) corticosteroids within 4 months prior to randomization or topical, rectal,or inhaled corticosteroids in current use more than 2 times per week.
12. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 3 years of the study.
13. Blood pressure greater than 180/110 (systolic above 180 or diastolic above 110).

    - If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.

    (Study Eye Inclusion Criteria:)

    The patient must have at least one eye meeting all of the inclusion criteria (a-d) and none of the exclusion criteria (e-x) listed.

    A patient may have two study eyes only if both are eligible at the time of randomization.

    The eligibility criteria for a study eye are as follows:
    1. Best corrected E-ETDRS visual acuity score of greater than or equal to 24 letters (i.e., 20/320 or better) and less than or equal to 68 letters (i.e., worse than 20/40).

       - There will be an enrollment limit of approximately 10% of eyes with visual acuity of 64 to 68 letters.
    2. Definite retinal thickening due to diabetic macular edema based on clinical exam involving the center of the macula.
    3. Mean retinal thickness on two OCT measurements greater than or equal to 250 microns in the central subfield.
    4. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs.

       (Study Eye Exclusion Criteria:)
    5. Macular edema is considered to be due to a cause other than diabetic macular edema.

       - An eye should not be considered eligible: (1) if the macular edema is considered to be related to cataract extraction or (2) clinical exam and/or OCT suggests that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema.
    6. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hare exudates, nonretinal condition).
    7. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
    8. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
    9. History of prior treatment with intravitreal corticosteroids.
    10. History of peribulbar steroid injection within 6 months prior to randomization.
    11. History of focal/grid macular photocoagulation within 15 weeks (3.5 months) prior to randomization.

        * Note: Patients are not required to have had prior macular photocoagulation to be enrolled.
        * Note: If prior macular photocoagulation has been performed, the investigator should believe that the patient may possibly benefit from additional photocoagulation.
    12. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization.
    13. Anticipated need for PRP in the 4 months following randomization.
    14. History of prior pars plana vitrectomy.
    15. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization.
    16. History of YAG capsulotomy performed within 2 months prior to randomization.
    17. Intraocular pressure greater than or equal to 25 mmHg.
    18. History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion).

        * A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is less than 25 mmHg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous.
        * Note: if the intraocular pressure is 22 to less than 25 mmHg, then the above criteria for ocular hypertension eligibility must be met.
    19. History of steroid-induced intraocular pressure elevation that required IOP-lowering treatment.
    20. History of prior herpetic ocular infection.
    21. Exam evidence of ocular toxoplasmosis.
    22. Aphakia.
    23. Exam evidence of pseudoexfoliation.
    24. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

    (Fellow Eye Inclusion Criteria:)

    In patients with only one eye meeting criteria to be a study eye at the time of randomization, the fellow eye must meet the following criteria:
    1. Best corrected E-ETDRS visual acuity score of greater than or equal to 19 letters (i.e., 20/400 or better).
    2. No prior treatment with intravitreal corticosteroids.
    3. Intraocular pressure less than 25 mmHg.
    4. No history of open-angle glaucoma (either primary open -angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion).

       * A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is less than 25 mmHg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous.
       * Note: if the intraocular pressure is 22 to less than 25 mmHg, then the above criteria for ocular hypertension eligibility must be met.
    5. No history of steroid-induced intraocular pressure elevation that required IOP-lowering treatment.
    6. No exam evidence of pseudoexfoliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2005-03-09; Study Completion 2006-10-30

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648